CLINICAL TRIAL: NCT02440048
Title: Using Boned-Apatite Cement at the Time of Extractions for Ridge Preservation at These Sites
Brief Title: Using Boned-Apatite Cement at the Time of Extraction for Ridge Preservation at These Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, machtei, Head - School of Graduate Dentistry & Chairman,Department of Periodontology, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0092-15-RMB CTIL; prof. Eli machtei (Other: Rambam Health Care Campus)
Record Dates: First submitted 2015-05-03; First posted 2015-05-12 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Alveolar Bone Loss
Keywords: extraction; Bond Apatite
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- HA ®Bond-apatite (Experimental): 10 extraction sockets will be preserved with Bond Apatite synthetic bone substitutes as test group
  Interventions: Device: Bond Apatite synthetic bone substitute
- BioOss bovine bone substitute (Active Comparator): 10 extraction sockets will be preserved with BioOss particles bovine bone substitute as a positive control
  Interventions: Device: BioOss bovine bone substitute
- extraction (No Intervention): 10 extraction sockets with no use of bone substitute as negative control.

INTERVENTIONS:
Device: Bond Apatite synthetic bone substitute — Synthetic bone grafts had been successful for ridge preservation. Calcium sulfate is the oldest material, being in use in dentistry for more than 30 years ago, and in orthopedics for more than 100 years ago. Calcium sulfate is completely absorbed and constitutes a matrix on wich bone is able to grow (osteoconductive). It does not induce inflammation and does not alter calcium levels in the blood flow.Previous studies has shown that calcium sulfate is completely replaced by bone. On the other hand, fast absorption of calcium sulfates can alter the dimensional stability of the graft. Adding Hydroxy Apatite may improve stability during bone remodeling.
  Arms: HA ®Bond-apatite
Device: BioOss bovine bone substitute — To assess efficiency of ridge preservation (in vertical and horizontal dimensions) after tooth extraction using Calcium Sulfate with HA (®Bond-apatite) compared to the use of bovine bone substitute (BioOss®) and to extraction only as negative control.
  Arms: BioOss bovine bone substitute

SUMMARY:
To assess efficiency of ridge preservation (in vertical and horizontal dimensions) after tooth extraction using Calcium Sulfate with hydroxyapatite(®Bond-apatite) compared to the use of bovine bone substitute (BioOss®) and to extration only as negative control.

DETAILED DESCRIPTION:
Dental implants have become in the past ten years a popular and promising treatment in the rehabilitation of missing teeth. However, using implants depends on adequate alveolar bone volume. Anatomical restrictions are mostly present in posterior mandibular and maxillary regions. Alveolar bone loss usually occurs because of active periodontal disease, trauma or teeth extractions.

Teeth extractions are associated with some loss of alveolar bone in the horizontal and vertical dimensions. This loss is more pronounced when teeth are extracted because of periodontal disease. Bone grafts from different origins (autogenic, allogenic, xenogenic or alloplastic) can partly reduce the alveolar bone loss. Different ridge preservation techniques were succesfully used in clinical trials, using membranes only or as a combination of membranes and bone substitutes.

Synthetic bone grafts have been proven successfully for ridge preservation. Calcium sulfate is the oldest material, being in use in dentistry for more than 30 years , and in orthopedics for more than 100 years . Calcium sulfate is completely absorbed and constitutes a matrix on wich bone is able to grow (osteoconductive). It does not induce inflammation and doesn't alter calcium levels in the blood flow.Previous studies has shown that calcium sulfate is completely replaced by bone. On the other hand, fast absorption of calcium sulfates can alter the dimensional stability of the graft. Adding Hydroxy Appatite may improve stability during bone remodeling.

This study includes patients who need extractions of incisors, canines or premolars. The extraction sockets must be mostly intact with a maximum 4 mm of one wall missing in the vertical dimension.

30 patients who need extractions from region of interest, with no extended bony defects, will be enrolled from the department of Periodontology, school of graduate dentistry, Rambam Health Care Campus

ELIGIBILITY:
Inclusion Criteria:

* Informed consent properly described and signed.
* Patients who need extractions of molars for dental or periodontal reasons.
* At least 18 years old.
* Need for future dental implants in the extraction areas.

Exclusion Criteria:

* No informed consent.
* Pregnant women.
* Women who breastfeed.
* Patients treated with drugs influencing metabolism of bone such as bisphosphonates.
* Heavy smokers (more than 20 cigarettes per day).
* Patients with dentures pressing on the area of extractions/bone grafts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
socket dimensions | 4 months
  Measurement of socket width (B-L aspect) in two vertical points and Distance from alveolar crest height in the middle of the socket to the marked point in the bottom of the stent.

SECONDARY OUTCOMES:
Complications | 4 month
  Complications will be documented: Infection, swelling, discomfort, pain, bone substitutes particles moving away from the tissue.

CONTACTS AND LOCATIONS:
Overall Officials: prof. Eli Machtei, DMD, Principal Investigator — Department of periodontology
Locations (1):
- Rambam Health Care Campus, Dept. of Periodontology, Haifa, Israel